CLINICAL TRIAL: NCT06391684
Title: Neurofunctional Specificities in Predictive Processing During High-Level Cognitive Flexibility Tasks in Autistic Males and Females
Brief Title: Flexibility and the Predictive Brain in Autistic Males and Females
Acronym: FLEX-PREAU
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0308; 2023-A01878-37 (Other: ID RCB)
Record Dates: First submitted 2024-02-08; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; flexibility; predictive coding; social cognition; sex differences
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autistic adults: Participants who have an autism diagnosis.
  Interventions: Behavioral: Social/non social; predictable vs unpredictable
- Non autistic adults: Participants who do not have an autism diagnosis
  Interventions: Behavioral: Social/non social; predictable vs unpredictable

INTERVENTIONS:
Behavioral: Social/non social; predictable vs unpredictable — Task 1: social predictable vs social unpredictable ; Task2 a. social & b. non social, predictable/unpredictable (for both)

SUMMARY:
The goal of this study is to compare the neural correlates of predictive brain mechanisms during high-level social and non-social flexibility tasks, between autistic and non-autistic males and females. The aim is to better understand if autistic individuals differ from non-autistic individuals in their cognitive flexibility according to the social and predictable nature of the stimuli, at a behavioral and neurofunctional level using the functional Magnetic Resonance Imaging (fMRI). As autistic females usually present a more subtle profile than autistic males, the investigators will also explore if autistic males and females present neurofunctional differences.

DETAILED DESCRIPTION:
Background:

Autism spectrum conditions (ASC) may involve specificities in predictive brain mechanisms, which guide perception together with sensory input. These predictive mechanisms are at play in various aspects of life, such as social interactions, in which autistic individuals have difficulties. They are also important for cognitive flexibility, which involves changing tasks, strategies, or perspectives according to the situation. recent research highlighted that autistic individuals faced difficulties in flexibly adjusting their predictions to unpredictable social contexts during a socio-emotional flexibility task (social stimuli). However, they found no difference between autistic and non-autistic individuals during a cognitive flexibility task involving predictable changes of non-social stimuli. This study aims to more precisely investigate which conditions lead to flexibility difficulties in autism (i.e., the social context, the unpredictability, or both) and to investigate the brain networks involved in autistic and non-autistic participants during high-level cognitive flexibility tasks involving social and non-social stimuli. In addition, autistic females often presenting better socio-communicational abilities than autistic males and a different profile from males in past research involving cognitive flexibility, the investigators will explore if they present a different neurofunctional signature from males during these tasks.

Procedure:

The protocol begins with an imaging localization phase (5 minutes). Subsequently, functional MRI tasks (T2*) commence. The protocol consists of two cognitive tasks, performed within the MRI scanner, each preceded by a training phase. The acquisition of each participant's anatomical sequence (T1; 5 minutes) is conducted between the first two cognitive tasks to avoid compromising participant concentration. Finally, functional connectivity data are collected during a 'resting state' sequence (10 minutes). The study comprises a single visit.

Cognitive Tasks:

The protocol starts with an Emotional Shifting Task (EST), where participants evaluate the valence of emotion (positive vs. negative) on an image while it's truncated; then, the image appears not truncated, and the participant must reevaluate its valence. In some cases, the valence has changed (from positive to negative or from negative to positive), and the participant must consider scene cues and demonstrate flexibility to reassess their judgment. This task lasts approximately 11 minutes.

In a second group of tasks, the participant will perform adapted versions of the Task-Switching Task (TST). In the first task, a letter and a number appear side by side, surrounded by either a blue or yellow frame. When the stimulus appears in a blue frame, the participant must focus on the letter and press the left response button if it's a consonant and the right response button if it's a vowel. When the stimulus appears in a yellow frame, the participant must focus on the numbers and press the left response button when it's odd and the right response button when it's even. In the first part, the subject first practices only the letter task to assimilate the task. Then, similarly, the subject practices only the number task. Finally, the subject performs the alternating task, with 2 conditions of predictability: predictable (task change every three trials), and not predictable (random change). This task lasts approximately 10 minutes. The second task adds an emotional component to the TST task: a face (male or female) associated with an emotion (positive or negative) is surrounded by either a blue or yellow frame. When the stimulus appears in a blue frame, the subject must focus on the gender and press the right response button if it's a female and the left response button if it's a male. When the stimulus appears in a yellow frame, the subject must focus on the facial emotion and press the right response button if it's a positive facial emotion and the left response button if it's a negative facial emotion. In the first part, the subject first practices only the gender task to assimilate the task. Then, similarly, the subject practices only the emotional task. Finally, the subject performs the alternating task, with the 2 conditions of predictability. This task also lasts 10 minutes.

Psychometric Assessment :

The subject will also undergo a psychometric assessment including the Social Responsiveness Scale (SRS), Camouflaging Autistic Trait - questionnaire (CAT-Q), Weschler Adult Intelligence Scale 4th edition (WAIS-4), Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A), Empathy Quotient (EQ), Autism Spectrum Quotient (AQ), and Autism Diagnostic Interview -revised (ADI-R) with the parent (if possible).

Hypotheses:

Given the literature, the investigators hypothesize a reduction in activation of certain areas in predictable conditions compared to unpredictable conditions, indicating the presence of a prediction error. Specifically, in the socio-emotional flexibility task (EST), the investigators expect to observe this reduction, particularly in the precuneus, the temporal lobe, the fusiform gyrus, and the locus coeruleus. In the cognitive flexibility task (adapted TST), the investigators will more specifically focus on the locus coeruleus. The investigators also anticipate observing the involvement of a global functional network showing differences in activations between autistic and non-autistic individuals, as well as a modulation of this reduction in activation (prediction error) between the two groups. Finally, the investigators hypothesize an intermediate profile in autistic females, both at the behavioral and neurofunctional level, situated between those of autistic males and non-autistic females.

Data Analysis:

Behavioral data will be analyzed in terms of accuracy rates and reaction times for both tasks. fMRI data will undergo classical analysis (General Linear Model - GLM). This GLM analysis will allow a direct comparison of experimental conditions within the same group of participants and identify possible differences in activations between the groups.

ELIGIBILITY:
Inclusion Criteria:

For non autistic individuals

* Affiliation with social security scheme.
* Registration in the national database of individuals willing to participate in research involving human subjects.
* Absence of contraindications for MRI.
* Signed informed consent before any study-related procedure.
* Visual acuity allowing normal perception of stimuli or corrected vision.
* Autism Quotient (AQ) (Baron-Cohen et al., 2001) < 32.

For autistic individuals:

* Affiliation with social security scheme.
* Absence of contraindications for MRI.
* Signed informed consent before any study-related procedure.
* Visual acuity allowing normal perception of stimuli or corrected vision.
* Diagnosis of autism established by a competent professional based on DSM/ICD criteria.

Exclusion Criteria:

* Any subject with a vascular stent implanted less than 6 weeks before the examination.
* Any subject with implanted biomedical material deemed "unsafe" or "not safe" in the list: http://www.mrisafety.com/TheList_search.asp.
* Any acquisition procedure not meeting the conditions required for "conditional" use in subjects with implanted biomedical material classified as "conditional" in the list: http://www.mrisafety.com/TheList_search.asp.
* Any subject with biomedical material such as a cardiac, neuronal, or sensory stimulator (cochlear implant due to the risk of demagnetization, heating, electrode, and artifacts) or a ventricular shunt valve without medical and paramedical supervision trained in MRI performance in these subjects.
* Intraocular or intracranial ferromagnetic foreign body near nerve structures (risk of displacement and complications such as ocular or cerebral lesions).
* Claustrophobia - Psychiatric or neurological conditions other than those specified.
* Existence of a severe general health condition incompatible with the study: cardiac, respiratory, hematological, renal, hepatic, or cancerous.
* Alcohol ingestion before the examination.
* Persons covered by articles L1121-5 to L1121-8 of the Public Health Code (pregnant or breastfeeding women, minors or adults under legal protection, individuals under administrative or judicial surveillance).
* Visual impairments.
* Intellectual disability.
* Inability to understand research instructions or provide informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Autistic with a diagnosis and non autistic adults.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Neurofunctional activity specificity of autistic adults in predictive processes during cognitive flexibility tasks | during activation tasks
  fMRI BOLD signal

SECONDARY OUTCOMES:
Functional connectivity specificity of autistic adults | through study completion, an average of 1 year
  BOLD-fMRI signal during resting state (BOLD-RS)
EST accuracy | through study completion, an average of 1 year
  the emotional shifting task (EST), is one of the task that will be performed in the fMRI. During this task participants evaluate the valence of emotion (positive vs. negative) on an image while it's truncated; then, the image appears not truncated, and the participant must reevaluate its valence. In some cases, the valence has changed (from positive to negative or from negative to positive), and the participant must consider scene cues and demonstrate flexibility to reassess their judgment.
  We will collect the accuracy of this task
EST response time | through study completion, an average of 1 year
  We will collect the response time in this task (described above)
TST accuracy | through study completion, an average of 1 year
  The Task-Switching Task (TST) is described in the study description. We will collect the accuracy of this task
TST response time | through study completion, an average of 1 year
  We will collect the response time in this task (described above)
SRS | through study completion, an average of 1 year
  The social responssivness scale is a scale giving a score between 0 and 195, that help to identify social difficulties in autism. Higher values indicate greater expression of the ASD-related phenotype. The self reported-version will be used.
AQ | through study completion, an average of 1 year
  The Autism spectrum quotient is a self-administrated questionnaire, with scores ranging from 0 to 50, that helps to identify autistic traits. Higher values indicate greater expression of the ASD-related phenotype
EQ | through study completion, an average of 1 year
  The empathy quotient is a self-administrated questionnaire, with scores ranging from 0 to 80. Higher values indicate high ability to understand how other people feel
CAT-Q | through study completion, an average of 1 year
  The Camouflaging Autistic Trait Questionnaire (CAT-Q) is a self-administered questionnaire, with scores ranging from 25 to 75. Higher values indicate greater camouflaging, i.e., greater ability to mask autistic symptoms in social contexts.
BRIEF-A | through study completion, an average of 1 year
  The Behavior Rating Inventory of Executive Function-Adult Version ( BRIEF-A) is a self-administrated questionnaire measuring executive dysfunctions. The global raw score can range from 70 to 210. Higher scores indicate greater executive dysfunctions
WAIS-IV | through study completion, an average of 1 year
  The Weschler Adult Intelligence Scale 4th edition (WAIS-IV) measure IQ. Higher scores indicate a higher Intelligence Quotient - IQ)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lacroix A, Dutheil F, Logemann A, Cserjesi R, Peyrin C, Biro B, Gomot M, Mermillod M. Flexibility in autism during unpredictable shifts of socio-emotional stimuli: Investigation of group and sex differences. Autism. 2022 Oct;26(7):1681-1697. doi: 10.1177/13623613211062776. Epub 2021 Dec 27. PMID 34957880